CLINICAL TRIAL: NCT03767023
Title: Clinical and Microbiological Relationships Between Periodontitis and Abdominal Aorta Aneurism: an Case Control Study
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Leila Salhi, Doctor of Dental Surgery (DDS), Master of sciences (MS), PhD student, University of Liege
Other Study IDs: H2014-3 AAA
Record Dates: First submitted 2018-10-26; First posted 2018-12-06 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Abdominal Aorta Aneurism; Periodontitis; Dentulous
MeSH Terms: conditions — Periodontitis | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — saliva, sub-gingival and supra-gingival samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stable AAA: = patients with a small abdominal aortic aneursym diameter < 55 mm "
  Interventions: Other: cross sectional
- instable AAA: =patients with a large abdominal aortic aneursym diameter > 55 mm and/or AAA with rapid growth who needs open surgery or EndoVascular Aneurysm Repair "EVAR
  Interventions: Other: cross sectional

INTERVENTIONS:
Other: cross sectional

SUMMARY:
Aorta Abdominal aneurism (AAA) is a chronic degenerative disorder leading to the dilation and eventually to the rupture of the aortic wall. The pathology presents risk factors such as aging, atherosclerosis, male gender, cigarette smoking, pulmonary emphysema and high blood pressure.The vascular wall destruction is characterized by a remodeling of the extracellular matrix (ECM), the presence of an inflammatory infiltrate of macrophages and lymphocytes associated increase in production of MMPs. A similar destruction mechanisms is found in periodontitis a chronic inflammatory diseases characterized by gram-negative bacteria species that are able to degrade ECM of the tooth supporting tissues and leading finally to tooth loss .Moreover, relationships between periodontitis and cardiovascular disease have already been demonstrated. These associations are considered to be initiated by transient or prolonged bacteremia due to dissemination of oral bacteria or their products into the bloodstream . The periopathogens, more specifically Porphyromonas gingivalis (Pg), were observed in atherosclerosis and aneurysm specimens as well as in coronary heart disease and endocarditis The association between periodontitis and Abdominal Aortic Aneurysms (AAA) has not often been studied especially from a clinical aspect. The mechanisms that induce the initiation, the development or the recurrence and the rupture of AAA after a period of quiescence not well studied and are therefore still unknown.

The aim of this clinical observational case controlled study is to search for a possible relationship between periodontal disease and rapid growth of AAA. Patients presenting stable or unstable AAA will be screened for the degree of periodontitis, for the type of oral microbiology and periodontopathogen markers present in the blood stream.

DETAILED DESCRIPTION:
31 consecutive dentulous patients diagnosed for AAA requiring a cardiovascular surgery (instable AAA) and 31 consecutive dentulous patients with stable AAA (no need for cardiovascular surgery) will be recruited from the Cardiovascular Surgery Department of the University Hospital of Liège (Faculty of Medicine, University of Liège, Belgium - Pr. N. Sakalihasan). The 62 patients will be subjected to:

1. Full clinical periodontal parameter assessment
2. Microbiological analyses of saliva,
3. Supra- and sub- gingival microbiological test
4. Blood test for biomarker analysis.
5. Imaging (echography, CT-Scans)measurments

ELIGIBILITY:
Inclusion Criteria:

* AAA
* dentulous
* ability to come in Hospital

Exclusion Criteria:

* diseases of connective tissue: rheumatoid arthritis, systemic lupus erythematosus, systemic sclerodermia, Crohn disease, Marfan syndrome, Heler Danlos syndrome, polymyosite/dermatomyosite, mix connectivite (MCDT)
* aneurysms of the lower limbs (femoral or popliteal)
* contraindication to the scanner
* participation of another clinical trial 30 days before baseline
* patient with risk oslerien
* taking antibiotics during the 3 months preceding the inclusion
* obese patients (BMI ≥ 30 kg/m2)
* immunosuppressant drugs or chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Cardiovascular Surgery Department, University Hospital of Liège (Belgium) and presenting AAA were screened in order to include 31 patients in each group (stable versus instable AAA) according to the sample size calculation. Sixty-two patients were therefore included according to the following inclusion and exclusion criteria:
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
pocked depth correlated with AAA stability | june 2017
  Periodontal clinical parameters such as pocked depth (PD, millimeter) will be correlated with AAA stability.

SECONDARY OUTCOMES:
pocked depth correlated with abdominal aortic aneurysm diametres such as anterior -posterior | March 2018
  Periodontal clinical parameters such as pocked depth (PD, millimeter) will be correlated with abdominal aortic aneurysm diametres such as anterior -posterior (AP,millimeter)